CLINICAL TRIAL: NCT02880306
Title: Hepatocellular Carcinoma and Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 05-W01-030
Record Dates: First submitted 2016-08-17; First posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- RA cohort: RA was diagnosed based on the 1987 American College of Rheumatology diagnostic criteria.
  Interventions: Other: RA
- Non-RA cohort: Participants who were ≥18 years of age, without a RA diagnosis

INTERVENTIONS:
Other: RA — RA was diagnosed based on the 1987 American College of Rheumatology diagnostic criteria
  Groups: RA cohort

SUMMARY:
Rheumatoid arthritis(RA) is a disorder with altered immunologic function and increased risk of developing malignancies, while studies examining the association between hepatocellular carcinoma (HCC) and RA remain lacking. The investigators aimed to investigate the risk of HCC between participants with and without RA.

DETAILED DESCRIPTION:
The investigators did a retrospective, observational, nested case-control study in a cohort that was previously recruited from a population-based RA survey. All participants were enrolled prospectively in Taiwan's national health insurance between Jan 1, 1999, and June 30, 2009, and had follow-up data until Dec 31, 2009. RA was diagnosed based on the 1987 American College of Rheumatology diagnostic criteria. The investigators matched RA and non-RA subjects by propensity score in a 1:1 ratio. The primary outcome was the risk of developing HCC. Cox proportional hazards regression was applied to estimate the hazard ratio (HR) and 95% confidence interval (CI) of HCC for RA and non-RA cohort.

ELIGIBILITY:
Inclusion Criteria:

* subjects were required to have ≥2 RA diagnosis (International Classification of Diseases, Ninth Revision [ICD-9-CM]-codes 714.0x), and to be ≥18 years of age on the date of first diagnosis. And inclusion in the Registry for Catastrophic Illness Patient Database (RCIPD)

Exclusion Criteria:

* who were diagnosed with RA only once during the study interval, <18 years of age when first diagnosed with RA, first diagnosed with RA after July 1, 2009, or not registered in the RCIPD were excluded

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All individuals were enrolled prospectively in Taiwan's national health insurance between Jan 1, 1999, and June 30, 2009, and had follow-up data until Dec 31, 2009
Sampling Method: Non-Probability Sample
Enrollment: 741379 (Actual)
Dates: Start 2014-07; Primary Completion 2016-03 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
the risk of developing hepatocellular carcinoma | between Jan 1, 1999 and Dec 31, 2009

IPD SHARING:
Plan to Share IPD: Yes
The Taiwan's National Health Insurance Research Database (NHIRD) between Jan 1, 1999, and June 30, 2009, and had follow-up data until Dec 31, 2009. The Taiwan's NHIRD contains health-care data gathered prospectively for 99% of Taiwan's population and approximately 22,600,000 individuals in 2007. The Taiwan's National Health Research Institutes (NHRI) maintained the NHIRD and provided it to the investigators for research purposes. De-identified data were further scrambled before being released to public access for research. The accuracy of diagnosis of major diseases in the NHIRD, such as stroke and acute coronary syndrome, has been validated previously.

REFERENCES:
- [Derived] Hsu CS, Lang HC, Huang KY, Chao YC, Chen CL. Risks of hepatocellular carcinoma and cirrhosis-associated complications in patients with rheumatoid arthritis: a 10-year population-based cohort study in Taiwan. Hepatol Int. 2018 Nov;12(6):531-543. doi: 10.1007/s12072-018-9905-7. Epub 2018 Nov 14. PMID 30426396